CLINICAL TRIAL: NCT01387100
Title: Efficacy of a Modified Vocational Rehabilitation Intervention for Work Disability
Brief Title: A Modified Rehabilitation Intervention for Working Persons With Arthritis
Acronym: Work It
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H133B100003-1
Record Dates: First submitted 2011-06-23; First posted 2011-07-04 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Arthritis
Keywords: supportive employment; vocational rehabilitation
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapist/Occupational Therapist Intervention (Experimental): This group will be assigned a physical therapist or occupational therapist to meet with followed by 2 phone consultations.
  Interventions: Behavioral: Vocational Rehabilitation Intervention
- Control (No Intervention): This is the control group. This group will not receive the vocational rehabilitation intervention from an occupational or physical therapist. They will receive written information regarding job accommodations and disability advocacy.

INTERVENTIONS:
Behavioral: Vocational Rehabilitation Intervention — Physical or occupational therapist will deliver a vocational rehabilitation intervention using the Work Experience Survey for Persons with Rheumatic Conditions (WES-RC) assessment tool to assess subject's health and vocational background as well as work barriers.
  Arms: Physical Therapist/Occupational Therapist Intervention

SUMMARY:
The purpose of this study is to explore the effects of a brief vocational rehabilitation intervention on individuals with arthritis who are concerned about their ability to remain employed.

ELIGIBILITY:
Inclusion Criteria:

* Live or work in eastern Massachusetts
* Age 25-63 years
* Risk of work loss due to arthritis
* Arthritis
* Chronic back pain
* Currently employed

Exclusion Criteria:

* Unemployed
* No arthritis

Ages: 25 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in work status | Baseline, 6, 12, 24 month follow up
  Work limitation will be assessed using the Work Limitation Questionnaire, a tool developed to assess limitation in ability to work due to health.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Keysor, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Sargent College of Health and Rehabilitation Sciences, Boston, Massachusetts, United States

REFERENCES:
- [Derived] AlHeresh R, Vaughan MW, Brenner IH, Keysor J. Recruitment cost and outcomes for an arthritis work disability prevention randomized clinical trial: The Work It study. Contemp Clin Trials Commun. 2021 Nov 12;24:100862. doi: 10.1016/j.conctc.2021.100862. eCollection 2021 Dec. PMID 34825102
- [Derived] Keysor JJ, LaValley MP, Brown C, Felson DT, AlHeresh RA, Vaughan MW, Yood R, Reed JI, Allaire SJ. Efficacy of a Work Disability Prevention Program for People with Rheumatic and Musculoskeletal Conditions: A Single-Blind Parallel-Arm Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Jul;70(7):1022-1029. doi: 10.1002/acr.23423. Epub 2018 Apr 25. PMID 28941189